CLINICAL TRIAL: NCT03003923
Title: A Randomised Control Trial of an Educational and Taste-exposure Intervention to Promote Vegetable Intake in Preschool Aged Children
Brief Title: Promoting Vegetable Intake in Preschool Aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Purely Nutrition Ltd (Unknown); Economic and Social Research Council, United Kingdom (Other)
Responsible Party: Principal Investigator, Chandani Nekitsing, Principal Investigator, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Chandani Nekitsing
Record Dates: First submitted 2016-12-15; First posted 2016-12-28 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Food Habits; Food Preferences; Behavior; Health Behavior
Keywords: Vegetable intake; Taste exposures; Educational intervention; Preschool children; Healthy eating intervention
MeSH Terms: conditions — Feeding Behavior; Food Preferences; Behavior; Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Taste Exposure (Experimental): Children will be repeatedly offered the single vegetable which is unfamiliar to them over the 12 week period. Children will be in their natural setting at nursery and will be offered 40g of the vegetable by their usual nursery staff. The vegetable will be weighed before and after using a digital scale by the researcher.
  Interventions: Behavioral: Taste exposure
- Nutritional Education (Experimental): Nursery staff will be trained by the PhunkyFoods team to deliver the nutritional education programme. Children will be taught Eat Well (learning about different food groups) and Strive for Five (learning about eating fruits and vegetables) components of the PhunkyFoods education programme by their usual nursery staff. Nurseries will be advised to deliver as much as possible of the two components over the 12 week period.
  Interventions: Behavioral: Nutritional education
- Taste Exposure and Nutritional Education (Experimental): Children will be repeatedly offered a single unfamiliar vegetable over the 12 week period as well as receive the PhunkyFoods educational programme (Eat Well and Strive for Five components). Children will be in their natural setting at nursery and will be offered the vegetable and nutritional education by their usual nursery staff.
  Interventions: Behavioral: Taste exposure; Behavioral: Nutritional education
- Control (No Intervention): Children will be offered single unfamiliar vegetable at the beginning, end and at the follow-up. There will be no repeated taste exposure or education during the study phase or follow-up; they will be offered the nutritional education after the study has completed.

INTERVENTIONS:
Behavioral: Taste exposure — Exposure to the same vegetable
  Arms: Taste Exposure; Taste Exposure and Nutritional Education
Behavioral: Nutritional education — Eat Well and Strive for Five nutritional education
  Arms: Nutritional Education; Taste Exposure and Nutritional Education

SUMMARY:
The aim of this cluster randomised control trial is to test the efficacy of a repeated taste exposure intervention, a nutritional educational intervention and combination of both to increase intake of an unfamiliar vegetable in preschool aged children (aged 3-5 years).

DETAILED DESCRIPTION:
The aim of this study is to test the efficacy of a repeated taste exposure intervention, a nutritional educational intervention and combination of both to increase intake of an unfamiliar vegetable in preschool aged children (aged 3-5 years). In particular the study will assess whether these strategies are effective to encourage intake of an unfamiliar vegetable in children who are fussy eaters or going through the food neophobia phase. The effectiveness of these interventions will also be observed overtime at 3 and 6 months post intervention.

Nurseries will be randomised into one of four conditions over the 12 week intervention period; these include educational intervention only, taste exposures only, taste exposures and educational intervention or no intervention (control group). All children will be offered an unfamiliar vegetable prior to the intervention and after the intervention to evaluate changes in intake of the unfamiliar vegetable. The repeated taste exposure groups will be offered the novel vegetable repeatedly (1 exposure per week) over the 12 week period. For the educational intervention nursery staff will be advised to deliver two components of an existing PhunkyFoods educational programme over the same period.

Parents will be asked some general demographic questions, child food behaviour questions and questions about their feeding practices. Finally nursery staff will be requested to provide feedback to evaluate intervention feasibility, barriers and efficacy.

It is predicted that children's intake of the unfamiliar vegetable will vary by intervention. The primary hypothesis to be tested is that children who receive the repeated taste exposures are more likely to increase their intake of the unfamiliar vegetable compared to those in educational only or control conditions. The second hypothesis is that repeated taste exposures will increase intake of an unfamiliar vegetable in fussy eaters more than education.

ELIGIBILITY:
Inclusion Criteria:

* 2 to 5 years old
* Attends nursery on selected test day

Exclusion Criteria:

* Relevant food allergy (mooli / radish)
* Medical condition which would prevent them from eating the test vegetable

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Intake of an unfamiliar vegetable | Week 0 (Pre Intervention Intake), Week 12 (Post Intake), Week 24 (Follow up 1), Week 36 (Follow up 2)
  Outcome measured at pre intervention (week 0), post intervention (week 12) and at follow-ups 3 (week 24) and 6 months (week 36) later. Intake of unfamiliar vegetable will be measured individually and objectively using weight in grams.

SECONDARY OUTCOMES:
Intake of usual vegetables | Week 0 (Pre Intervention Intake), Week 12 (Post Intake), Week 24 (Follow up 1)
  Outcome measured at pre intervention (week 0), post intervention (week 12) and at follow-up 3 months later (week 24). Intake of usual vegetable will be measured using a Food Frequency Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Chandani Nekitsing, MSc, Principal Investigator — University of Leeds
Locations (1):
- School of Psychology, University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No